CLINICAL TRIAL: NCT03697811
Title: An Open-Label, Multicenter Study Assessing the Efficacy and Safety of DE-117 Ophthalmic Solution 0.002% in Latanoprost Low/Non-Responder Subjects Diagnosed With Primary Open-Angle Glaucoma or Ocular Hypertension - Spectrum 5 Study
Brief Title: DE-117 Spectrum 5 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 011711IN
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Primary Open-angle Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DE-117 Ophthalmic Solution 0.002% (Experimental): Interventional treatment will be made with DE-117 Ophthalmic Solution 0.002% once daily in the evening for the duration of the 3 month treatment period.
  Interventions: Drug: DE-117 Ophthalmic Solution

INTERVENTIONS:
Drug: DE-117 Ophthalmic Solution — Interventional treatment will be made with DE-117 Ophthalmic Solution 0.002% once daily in the evening for the duration of the 3 month treatment period.

SUMMARY:
Santen will evaluate the intraocular pressure (IOP) lowering effect and efficacy of DE-117 ophthalmic solution 0.002% in latanoprost low/non-responder subjects diagnosed with POAG or OHT

ELIGIBILITY:
Inclusion Criteria:

* Patients with Primary Open-Angle Glaucoma or Ocular Hypertension in one or both eyes.
* Provide signed written informed consent.
* Diagnosis of POAG or OHT in both eyes.
* Qualifying corrected visual acuity in each eye.
* Qualifying central corneal thickness in each eye.
* Qualifying Day 1 IOP measurement at 3 time-points in both eyes after latanoprost Run-in Period.
* Qualifying Anterior chamber angle.
* Qualifying IOP measurement at 3 time-points during latanoprost Run-in Period.

Exclusion Criteria:

* Patients who cannot safely discontinue use of Ocular Hypotensive Medications during Washout.
* Patients with prior exposure to DE-117.
* History of ocular surgery specifically intended to lower IOP
* Advanced glaucoma in either eye.
* Any corneal abnormality or other condition interfering with or preventing reliable Goldmann applanation tonometry.
* Any ocular surgery or ocular laser treatment within 180 days prior to Visit 1 (Screening) and throughout the study in either eye.
* Females who are pregnant, nursing, or planning a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Arizona Eye Center, Chandler, Arizona
  - Global Research Management, Glendale, California
  - North Valley Eye Medical Group, Mission Hills, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Danbury Eye Physicians & Surgeons, Danbury, Connecticut
  - Shettle Eye Research, Inc., Largo, Florida
  - International Eye Associates, PA, Ormond Beach, Florida
  - Dixon Eye Care, Albany, Georgia
  - Clayton Eye Clinical Research, LLC, Morrow, Georgia
  - Coastal Research Associates, LEC, Roswell, Georgia
  - Heart of America Eye Care, P.A., Shawnee Mission, Kansas
  - Tekwani Vision Center, St Louis, Missouri
  - Comprehensive Eye Care Ltd, Washington, Missouri
  - NYU Langone Health Department of Ophthalmology, New York, New York
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - South Shore Eye Center, Wantagh, New York
  - Asheville Eye Associates, PLLC, Asheville, North Carolina
  - Mundorf Eye Center, Charlotte, North Carolina
  - Cornerstone Health Care, High Point, North Carolina
  - Apex Eye Clinical Research, LLC, Cincinnati, Ohio
  - Abrams Eye Center, Cleveland, Ohio
  - The Eye Institute, Tulsa, Oklahoma
  - Scott & Christie and Associates PC, Cranberry Township, Pennsylvania
  - Glaucoma Consultants and Center for Eye Research, PA, Mt. Pleasant, South Carolina
  - Total Eye Care PA, Memphis, Tennessee
  - VRF Eye Specialty Group, Memphis, Tennessee
  - Nashville Vision Associates, Nashville, Tennessee
  - Texas Eye, PA, Austin, Texas
  - Eye Clinic of Texas, League City, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas

REFERENCES:
- [Derived] Panarelli JF, Bowden EC, Tepedino ME, Odani-Kawabata N, Pei Z, McLaurin EB, Ropo A. Omidenepag Isopropyl in Latanoprost Low/Nonresponders With Primary Open Angle Glaucoma or Ocular Hypertension: A Phase 3, Nonrandomized, Two-Phase, Open-Label Study. J Glaucoma. 2023 Dec 1;32(12):999-1005. doi: 10.1097/IJG.0000000000002321. Epub 2023 Oct 17. PMID 37853676

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DE-117 Ophthalmic Solution 0.002%
Started | 107
Completed | 104
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | DE-117 Ophthalmic Solution 0.002%
Number analyzed (Participants) | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 91
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 42
  White | 64
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 107

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Diurnal Intraocular Pressure (IOP) at Month 3.
Description: IOP lowering effect of DE-117 ophthalmic solution 0.002% in Latanoprost low/non-responder subjects. Mean Diurnal Intraocular Pressure: Analysis of Change from Baseline in IOP score at Month 3 using Paired T-test on Observed Case. Mean Diurnal IOP is defined as the average IOP of all three timepoints (8:00,12:00, 16:00) at Month 3.
Time Frame: Month 3
Population: Full Analysis Set (observed cases only)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002%
Number analyzed (Participants) | 102
mmHg | -2.96 (2.831)

2. Secondary Outcome: Percent Change From Baseline in Mean Diurnal IOP at Week 2, Week 6 and Month 3
Description: The secondary efficacy endpoint evaluated percent change from baseline in mean DIOP at week 2, 6 and month 3.
Time Frame: week 2, 6 and month 3
Population: Full Analysis Set (observed cases only).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DE-117 Ophthalmic Solution 0.002%
Number analyzed (Participants) | 107
Percent change
  Week 2: number analyzed (Participants) | 105
  Week 2 | -12.21 (10.855)
  Week 6: number analyzed (Participants) | 106
  Week 6 | -12.40 (11.218)
  Month 3: number analyzed (Participants) | 102
  Month 3 | -12.57 (11.907)

3. Secondary Outcome: Change From Baseline in Mean Diurnal IOP at Week 2 and Week 6
Description: Change from baseline (Visit 4) in mean diurnal IOP at Week 2 (Visit 5) and Week 6 (Visit 6).
Time Frame: week 2 and 6
Population: Full Analysis Set (observed cases only).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002%
Number analyzed (Participants) | 107
mmHg
  Week 2: number analyzed (Participants) | 105
  Week 2 | -2.87 (2.531)
  Week 6: number analyzed (Participants) | 106
  Week 6 | -2.89 (2.578)

4. Secondary Outcome: Change From Baseline in IOP at Timepoints at Week 2
Description: Change in mean IOP were evaluated at each time point at all post-baseline visits. (Change from baseline measurement at each timepoint was calculated by deducting the baseline value at corresponding timepoint from the IOP measurement).
Time Frame: 08:00, 12:00 and 16:00 at Week 2
Population: Full Analysis Set (observed cases only).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002%
Number analyzed (Participants) | 107
mmHg
  8:00: number analyzed (Participants) | 105
  8:00 | -2.52 (2.976)
  12:00: number analyzed (Participants) | 105
  12:00 | -2.94 (2.922)
  16:00: number analyzed (Participants) | 105
  16:00 | -3.15 (3.077)

5. Secondary Outcome: Change From Baseline in IOP at Timepoints at Week 6
Description: Change in mean IOP were evaluated at each time point at all post-baseline visits.
Time Frame: 08:00, 12:00 and 16:00 at Week 6
Population: Full Analysis Set (observed cases only)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002%
Number analyzed (Participants) | 107
mmHg
  8:00: number analyzed (Participants) | 106
  8:00 | -2.42 (3.209)
  12:00 | -2.86 (2.832)
  16:00 | -3.44 (3.127)

6. Secondary Outcome: Change From Baseline in IOP at Timepoints at Month 3
Description: Change in mean IOP were evaluated at each time point at all post-baseline visits.
Time Frame: 08:00, 12:00 and 16:00 at month 3
Population: Full Analysis Set (observed cases only).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002%
Number analyzed (Participants) | 107
mmHg
  8:00: number analyzed (Participants) | 103
  8:00 | -2.76 (3.180)
  12:00: number analyzed (Participants) | 102
  12:00 | -2.98 (3.200)
  16:00: number analyzed (Participants) | 103
  16:00 | -3.08 (3.186)

7. Secondary Outcome: Intraocular Pressure: Percent Change From Baseline by Analysis Visit and Timepoint at Week 2
Description: Intraocular Pressure: Percent Change from Baseline by Analysis Visit and Timepoint.
Time Frame: 08:00, 12:00 and 16:00 at week 2
Population: Full Analysis Set (observed cases only).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DE-117 Ophthalmic Solution 0.002%
Number analyzed (Participants) | 107
Percent change
  8:00: number analyzed (Participants) | 105
  8:00 | -10.42 (12.509)
  12:00: number analyzed (Participants) | 105
  12:00 | -12.51 (12.765)
  16:00: number analyzed (Participants) | 105
  16:00 | -13.47 (13.204)

8. Secondary Outcome: Intraocular Pressure: Percent Change From Baseline by Analysis Visit and Timepoint at Week 6
Description: Intraocular Pressure: Percent Change from Baseline by Analysis Visit and Timepoint.
Time Frame: 08:00, 12:00 and 16:00 at week 6
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DE-117 Ophthalmic Solution 0.002%
Number analyzed (Participants) | 107
Percent change
  8:00: number analyzed (Participants) | 106
  8:00 | -10.04 (13.653)
  12:00 | -12.22 (12.432)
  16:00 | -14.80 (13.482)

9. Secondary Outcome: Intraocular Pressure: Percent Change From Baseline by Analysis Visit and Timepoint at Month 3
Description: Intraocular Pressure: Percent Change from Baseline by Analysis Visit and Timepoint.
Time Frame: 08:00, 12:00 and 16:00 at month 3.
Population: Full Analysis Set (observed cases only).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DE-117 Ophthalmic Solution 0.002%
Number analyzed (Participants) | 107
Percent change
  8:00: number analyzed (Participants) | 103
  8:00 | -11.43 (13.133)
  12:00: number analyzed (Participants) | 102
  12:00 | -12.72 (13.467)
  16:00: number analyzed (Participants) | 103
  16:00 | -13.13 (13.309)

ADVERSE EVENTS:
Time Frame: Adverse events in this study were collected from the time of informed consent and were followed to resolution, or until the subject's participation in the study ended at Month 3.
Description: Adverse events (AEs) are presented for the Safety analysis population. AEs were defined as any untoward medical occurrence in the study irrespective of a causal relationship with the study medication. AEs were followed to resolution and until the subject's exit from the study.
Arm/Group | DE-117 Ophthalmic Solution 0.002%
All-Cause Mortality (participants affected / at risk) | 0/107
Serious Adverse Events (participants affected / at risk) | 0/107
Other Adverse Events (participants affected / at risk) | 27/107
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DE-117 Ophthalmic Solution 0.002% (N=107)
Eye pain (Eye disorders) | 2
Anterior chamber cell (Eye disorders) | 1
Conjunctival oedema (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eyelash hyperpigmentation (Eye disorders) | 1
Macular oedema (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Instillation site foreign body sensation (General disorders) | 1
Instillation site pain (General disorders) | 1
Suture related complication (Injury, poisoning and procedural complications) | 1
Vital dye staining cornea present (Investigations) | 1
Bronchitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Cyst (General disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 9
Punctate keratitis (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT03697811/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT03697811/SAP_001.pdf